CLINICAL TRIAL: NCT01480583
Title: A Phase II, Multi-center, Open-label Study Evaluating GRN1005 Alone or in Combination With Trastuzumab in Breast Cancer Patients With Brain Metastases
Brief Title: GRN1005 Alone or in Combination With Trastuzumab in Breast Cancer Patients With Brain Metastases
Acronym: GRABM-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Angiochem Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP1005B016
Record Dates: First submitted 2011-11-16; First posted 2011-11-29 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Brain Metastases
Keywords: GRN1005; ANG1005; Peptide-Drug Conjugate (PDC); LRP-1; Targeted Therapy; Breast Cancer; Brain Metastases; Brain Tumor; Blood Brain Barrier; Trastuzumab; Herceptin; Paclitaxel; Taxol; Breast cancer with brain metastases
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — paclitaxel-Angiopep-2 conjugate; Trastuzumab; alovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GRN1005 (Experimental): GRN1005 alone in HER2- MBC patients with brain mets. 18F-FLT may also be administered to this arm (if patient enrolled at NCI)
  Interventions: Drug: GRN1005; Drug: 18F-FLT
- GRN1005 with trastuzumab (Experimental): GRN1005 in combination with trastuzumab in MBC patients with brain mets 18F-FLT may also be administered to this arm (if patient enrolled at NCI)
  Interventions: Drug: GRN1005; Drug: Trastuzumab; Drug: 18F-FLT

INTERVENTIONS:
Drug: GRN1005 — 550 mg/m2 IV every 3 weeks
  Other Names: ANG1005
Drug: Trastuzumab — 2 mg/kg IV every week or 6 mg/kg IV every 3 weeks per investigator choice
  Other Names: Herceptin
  Arms: GRN1005 with trastuzumab
Drug: 18F-FLT — 5 mCi of 18F-FLT IV during Screening and during Cycle 1
  Other Names: 18F-fluorothymidine

SUMMARY:
The purpose of this study is to assess the efficacy, safety, and tolerability of GRN1005 in patients with brain metastases from breast cancer. For patients with HER2 positive metastatic breast cancer, GRN1005 will be assessed in combination with Trastuzumab (Herceptin®) as per standard-of-care practice.

In addition, this study will evaluate the ability of 18F-FLT to determine if the amount of change in the uptake in the brain metastases from breast cancer after GRN1005 treatment, correlates with intra-cranial response (for patients enrolled at NCI).

DETAILED DESCRIPTION:
Please see Brief Summary section.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically or cytologically-documented breast cancer (HER2 status and ER/PgR status must be known)
3. Brain metastasis from breast cancer with or without prior WBRT
4. At least one radiologically-confirmed and measurable metastatic brain lesion (≥ 1.0 cm in the longest diameter) by Gd-MRI of the brain < 14 days prior to first dose (Metastatic brain lesions previously treated with SRS may not be target or non-target lesions)
5. Patients must be neurologically stable: On stable doses of corticosteroids and anticonvulsants (not EIAEDs, including phenytoin, phenobarbitol, carbamazepine, fosphenytoin, primidone, oxcarbazepine) for ≥ 5 days prior to obtaining the baseline Gd-MRI of the brain and ≥ 5 days prior to first dose
6. KPS ≥ 70%
7. Completed WBRT for intra-cranial lesions ≥ 28 days prior to first dose

Key Exclusion Criteria:

1. NCI CTCAE v4.0 Grade ≥ 2 neuropathy
2. CNS disease requiring immediate neurosurgical intervention (e.g., resection, shunt placement, etc.)
3. Known leptomeningeal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Intra-cranial objective response rate in breast cancer patients with brain metastasis | Upon enrollment through end of study period (1 year after last patient is enrolled)

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability of GRN1005 alone or in combination with Trastuzumab | Upon enrollment through end of study period (1 year after last patient is enrolled)
Intra-cranial objective response duration | Upon enrollment through end of study period (1 year after last patient is enrolled)
3-month intra-cranial progression-free survival | Upon enrollment through end of study period (1 year after last patient is enrolled)
Six month overall survival (OS) | Upon enrollment through end of study period (1 year after last patient is enrolled)

CONTACTS AND LOCATIONS:
Overall Officials: Betty Lawrence, Study Director — Angiochem Inc; Nancy Lin, MD, Principal Investigator — Dana-Farber Cancer Institute; Susan Bates, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Ingalls Memorial Hospital, Harvey, Illinois
  - NCI, Rockville, Maryland